CLINICAL TRIAL: NCT02084849
Title: The Autosomal Dominant Polycystic Kidney Disease (ADPKD) Cohort Study
Brief Title: ADPKD Cohort Study
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: PKD Foundation (Other)
Responsible Party: Principal Investigator, Arlene Chapman, Principal Investigator, Emory University
Other Study IDs: IRB00041117; 0247-1998 (Other: Other)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 84 Months
Biospecimen Retention: Samples With DNA — Whole blood, serum, urine, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Group 1 will consist of 300 ADPKD individuals who are early in the course of their disease and demonstrate risk factors for progression to ESRD.
- Group 2: Group 2 will consist of ADPKD subjects who have progressed to a more advanced stage of their renal disease. There is no limit with regard to the number of subjects to be recruited into this group.

SUMMARY:
The purpose of this study is to find out if radiology tests of the kidneys as opposed to glomerular filtration (GFR) tests (GFR test - a lab test that measures kidney function) follow progression of polycystic kidney disease (PKD) the best. PKD patients at risk for progression to renal failure (dialysis or transplantation) have been identified and include those who have been diagnosed with high blood pressure early, the presence of the PKD1 gene (the inherited abnormality responsible for the majority of PKD), men as opposed to women, those with episodes of visible blood or increased protein in their urine, and women who have experience more than three pregnancies. Individuals who are diagnosed with PKD in the first year of life or in utero (before birth) are also at high risk for progression to renal failure.

This study will also facilitate understanding of human diseases at the cellular and molecular level. We will be identifying genetic factors that may influence the severity of polycystic kidney disease (PKD). You are being asked to provide a sample of blood for the purpose of DNA or other biochemical analyses.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Hypertension diagnosed early in the course of the disease (less than 25 years for men; less than 30 years for women)
* ADPKD diagnosed in utero or in the first year of life
* The presence of proteinuria (between 180 mg and 1 gm/day) without evidence of a second renal disorder
* A history of more than 3 pregnancies and hypertension
* A history of gross hematuria
* A serum creatinine concentration less than 1.4 mg/dl
* ADPKD diagnosed in childhood with more than 10 cysts

Group 2

* Serum creatinine concentration >1.4 and
* Renal length greater than 15 cm and
* Age less than 60 years of age
* Severe pain or discomfort as assessed by the primary care physician related to ADPKD

Exclusion Criteria:

* Subjects, who in the assessment of the principal investigator cannot provide reliable follow-up
* Subjects who cannot be exposed to iothalamate
* Subjects who cannot undergo MRI due to the presence of a pacemaker or surgical clip in the abdomen
* Subjects who are not anticipated to survive during the duration of the study (e.g. underlying malignancy)
* Subjects who cannot provide informed consent
* Women who are pregnant or who have undergone a pregnancy in the last 6 months or who are presently breastfeeding

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: ADPKD individuals at risk for progression to End Stage Renal Disease (ESRD)
Sampling Method: Non-Probability Sample
Enrollment: 624 (Actual)
Dates: Start 1998-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in GFR as compared to change in renal volume over time | Three years

SECONDARY OUTCOMES:
Differences in the ability to determine change in renal volume over time between MRI and ultrasound | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Chapman, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States